## Statistical analysis

Statistical for Health Sciences Package Analysis (SPSS) will be performed using version 22.0 software (SPSS Inc., Chicago, IL, USA). Descriptive statistics, mean, standard deviation, or percentages will be collected. The significance level will be accepted as p  $\leq$ 0.005. The normality of the data will be evaluated using the Shapiro-Wilk test.

A Chi-square test will compare categorical (nominal) variables between groups. Continuous variables will be compared with the T-test when there are parametric samples between two groups or the Mann-Whitney U test when the models are not parametric. Results will be analyzed using a two-factor repeated measure analysis of variance followed by post-hoc tests. The significance level of the study, P: 0.05 value and 95% confidence interval (CI), will be considered statistically significant.